CLINICAL TRIAL: NCT05068024
Title: A Phase 1/2, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-Tumor Activity of FWD1509 MsOH in Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of FWD1509 in Adults With Non-Small Cell Lung Cancer
Acronym: FWD1509
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Forward Pharmaceuticals Co., Ltd. (Industry)
Collaborators: WuXi Clinical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWDCT-001
Record Dates: First submitted 2021-09-14; First posted 2021-10-05 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: FWD1509 MsOH in advanced non-small cell lung cancer; Forward Pharma; Forward; FWD1509; NSCLC; MsOH; FWD-001; First-in-human; Non-small cell lung cancer; Advanced solid malignancies; Solid malignancies; Solid tumor; EGFR; EGFR ex20ins; EGFR mutation; TKI; HER2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment of NSCLC patients with EGFR or HER2 genetic alterations (Experimental)
  Interventions: Drug: FWD1509 MsOH

INTERVENTIONS:
Drug: FWD1509 MsOH — FWD1509 MsOH is administered orally once daily. The starting dose is 10 mg/day for dose-escalation phase, and the dose level to be investigated in the expansion study will depend on the emerging data. For dose-extension phase, the recommended Phase 2 dose will be administered.

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of FWD1509 MsOH in advanced NSCLC patients and establish the maximum tolerable dose (MTD), recommended phase 2 dose (RP2D) in advanced NSCLC patients.

DETAILED DESCRIPTION:
This study will be a first-in-human study evaluating the safety and tolerability of FWD1509 MsOH in subjects with advanced NSCLC, when FWD1509 MsOH is administered once daily as a single agent. FWD1509 MsOH is an oral TKI (Tyrosine Kinase Inhibitor) that blocks the function of tyrosine kinase. TKIs such as gefitinib, erlotinib or afatinib are recommended as the first-line therapy for EGFR mutated (exon 19 deletions or L858R point mutations in exon 21) NSCLC patients. However, the majority (>50%) of patients will develop acquired resistance after initially responding to gefitinib or erlotinib due to the occurrence of secondary mutations (mostly T709M) in EGFR. Osimertinib was subsequently developed to such secondary mutations, but for EGFRex20ins mutations, on which there is still no effective therapies focusing. FWD1509 MsOH is new generation EGFR-TKI targeting EGFR mutations such as exon 19 deletion, L858R substitution as well as T790M mutations. In particular, FWD1509 MsOH targets the EGFRex20ins mutation in NSCLC. In addition to activity against EGFR mutations, FWD1509 MsOH is also active against a variety of HER2 mutations.

The development of FWD1509 MsOH at this stage is mainly focused on treatment of NSCLC tumors with EGFRex20ins mutations, followed by further exploration against other targets.

ELIGIBILITY:
Key Inclusion Criteria: Study-Wide Eligibility (Across All Study Parts):

A subject will be eligible for inclusion in this study only if all of the following criteria apply.

1. Have histologically or cytologically confirmed locally advanced or metastatic NSCLC (Stage IIIB/IIIC or IV) [JACC edition 8], and inclusion of Stage IIIB only if not a candidate for curative therapy
2. Must have sufficient tumor tissue (either archived sample or recent biopsy) available for analysis:

   1. Phase 1 Dose-escalation part: EGFR and HER2 mutations (including but not limited toL858R, exon 19 deletion, T790M, ex20ins, 21exon, G719X, S768I, L861Q, etc. for EGFR and A775YVMG, C776insVC, P780ins GSP etc. for HER2) should be confirmed by previously documented evidence or central lab
   2. Patients with both EGFR and HER2 mutations may be included in the dose escalation phase
   3. Phase 1 Dose-expansion part and Phase 2: Have an EGFR in-frame exon 20 insertion test by any central lab
3. Must have at least one measurable lesion as defined by response evaluation criteria in solid tumors (RECIST v1.1)
4. Prior anti-cancer therapies:

   1. Previously treated with one or more regimens of systemic therapy for locally advanced or metastatic disease
   2. Disease progressed or intolerant to at least one line of systematic therapies including but not limited to any EGFR-target therapies or immunotherapies, for metastatic / local relapsed settings
5. Male or female adult participants (aged 18 years or older, or as defined per local regulations)
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
7. Minimum life expectancy of 3 months or more
8. Adequate organ function at baseline

   1. Bone marrow function

      * Absolute neutrophil count (ANC)≥1.5 x 10^9/L
      * Platelets ≥100 x 10^9/L
      * Hemoglobin ≥9 g/dL, criteria must be met without a transfusion within 2 weeks of the blood draw
   2. Hepatic function

      * AST and ALT ≤3 x upper limit of normal (ULN); if liver metastases, then ≤ 5 x ULN
      * Bilirubin ≤1.5 x ULN or ≤3 x ULN in the presence of documented Gilbert's Syndrome
   3. Renal function

      * Creatinine clearance ≥50 ml/min (calculated by Cockcroft and Gault equation (Cockcroft DW, 1976) (Appendix 3)
9. Willingness and ability to comply with scheduled visits and study procedures

Exclusion Criteria:

A subject will be not eligible for inclusion in this study if any of the following criteria apply:

1. Received anticancer therapy including cytotoxic chemotherapy, biological products and investigational agents, ≤ 21 days prior to first dose of FWD1509 MsOH; or received prior EGFR TKIs (e.g., gefitinib, erlotinib or osimertinib) ≤7 days prior to the first dose FWD1509 MsOH
2. Have been diagnosed with another primary malignancy other than NSCLC except for patients with adequately treated non-melanoma skin cancer, cervical cancer in situ or definitively treated non-metastatic prostate cancer, or participants with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy
3. Received radiotherapy ≤14 days prior to the first dose of FWD1509 MsOH or have not recovered from radiotherapy-related toxicities; palliative radiation administered outside the chest and brain, stereotactic radiosurgery (SRS), and stereotactic body radiotherapy are allowed up to 7 days prior to the first dose of FWD1509 MsOH
4. Received strong CYP3A inhibitors and inducers within 2 weeks prior to the first dose of FWD1509 MsOH; they should be discontinued at least 2 weeks prior to the first dose of FWD1509 MsOH and avoided throughout the study duration (see Appendix 6)
5. Received concomitant medications (e.g., statins) which are substrates of BCRP, p-glycoprotein or OATP1B1/1B3 (dose escalation part of phase 1 study)
6. Have undergone major surgery within 28 days prior to first dose of FWD1509 MsOH. Minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed
7. Brain Metastasis: Have known active brain metastases (have either previously untreated intracranial CNS metastases or previously treated intracranial CNS metastases with radiologically documented new or progressing CNS lesions), except for the following conditions

   1. Brain metastases are allowed if they have been treated with surgery and/or radiation and have been stable without requiring corticosteroids to control symptoms within 7 days before the first dose of FWD1509 MsOH and have no evidence of new or enlarging brain metastases
   2. Requiring corticosteroids to control symptoms within 7 days prior to the first dose of FWD1509 MsOH or during study period; patients previously treated for CNS metastases who are clinically stable, have no new lesions, and who do not need treatment with a corticosteroid within the 7 days before the first dose of FWD1509 MsOH and during study period are allowed to be enrolled
8. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging) or leptomeningeal disease (symptomatic or asymptomatic)
9. Have significant, uncontrolled, or active cardiovascular disease
10. QCc-related criteria:

    1. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1) using Fredericia's QT correction formula
    2. A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome
11. Have significant, uncontrolled, or active renal disease
12. Have a known history of uncontrolled hypertension (per institution practice); participants with hypertension should be under treatment on study entry to control blood pressure
13. Have any abnormal changes in the cornea or retina that may increase the risk of ocular toxicity during screening
14. Have an ongoing or active infection, including but not limited to, the requirement for intravenous (IV) antibiotics, or a known history of human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Testing is not required in the absence of history
15. Currently have or have a history of interstitial lung disease, radiation pneumonitis that required steroid treatment, or drug-related pneumonitis
16. Female participants who are lactating and breastfeeding or have a positive urine or serum pregnancy test during the screening period
17. Have gastrointestinal illness or disorder that could affect oral absorption of FWD1509 MsOH
18. Have any condition or illness that, in the opinion of the investigator, might compromise participant safety or interfere with the evaluation of the safety of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
22-30 participants with treatment-related adverse events as assessed based on CTCAE v5.0. | 18 months
  Adverse events (AE), serious adverse events (SAE) and adverse events of special interest (AESI) will be assessed by Common Terminology Criteria for Adverse Events (CTCAE 5.0) grading system, changing from baseline and each treatment cycle (1 cycle=3 weeks). An Adverse Event (AE) is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for FWD1509 MsOH | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for FWD1509 MsOH | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
T1/2: Terminal Half-life for FWD1509 MsOH | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
  Terminal plasma half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, and not the time required to eliminate half the administered dose.
AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to infinite time for FWD1509 MsOH | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for FWD1509 MsOH | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
AUC0-24: Area Under the Plasma Concentration versus Time Curve From Time 0 to Time 24h for FWD1509 | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
AUCss: Area Under the Plasma Concentration versus Time Curve From Time 0 to the End of the Dosing Interval | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Apparent Plasma Clearance (CL/F), Apparent Volume of Distribution and Mean Residence Time (MRT) | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Extent of Accumulation on Multiple Dosing (Rac) | Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
ORR: Objective Response Rate | 18 months
  Confirmed ORR is defined as the proportion of participants who are confirmed to have achieved complete response (CR) or partial response (PR).
DoR: Duration of Response | 18 months
  Duration of response is defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that PD is objectively documented.
DCR: Disease Control Rate | 18 months
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) (in the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks) after the initiation of study drug.
PFS: Progression Free Survival | 18 months
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for progressive disease (PD) according to RECIST version 1.1 are met or death, whichever occurs first.
OS: Overall Survival | 18 months
  OS is defined as the interval from the date of randomization until death.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Gabrail Cancer Center, Canton, Ohio
  - MD Anderson Cancer Center, Houston, Texas